CLINICAL TRIAL: NCT05157516
Title: Ultrasound-Guided Lumbar Erector Spinae Plane Block Versus Caudal Block for Postoperative Analgesia in Hip and Proximal Femur Surgery in Pediatric Patients: A Prospective Randomized Controlled Study
Brief Title: Ultrasound-Guided Lumbar Erector Spinae Plane Block Versus Caudal Block for Postoperative Analgesia in Hip and Proximal Femur Surgery in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-340-2020
Record Dates: First submitted 2021-09-28; First posted 2021-12-15 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group ESPB (Active Comparator): Erector Spinae Plane Block
  Interventions: Procedure: erector spinea block
- In group CEA (Active Comparator): Caudal epidural block
  Interventions: Procedure: Caudal epidural block

INTERVENTIONS:
Procedure: erector spinea block — the patients will receive a single injection erector spinea block after induction of general anesthesia
  Arms: group ESPB
Procedure: Caudal epidural block — the patients will receive caudal epidural block after induction of general anesthesia
  Arms: In group CEA

SUMMARY:
The study will compare Ultrasound-Guided Lumbar Erector Spinae Plane Block and caudal block for Postoperative Analgesia in Hip and Proximal Femur Surgery in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.
* Scheduled to undergo hip or proximal femur surgeries.

Exclusion Criteria:

* Refusal of participation by parents or caregivers
* Known local anesthetic (LA) drug sensitivity
* Bleeding disorders with INR > 1.5 and/or platelets < 100,000/mm3.
* Skin lesions or wounds at the site of proposed needle insertion.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Pain score | 2 hours post-operatively
  By using face, legs, activity, and cry consolability scale [FLACC ]
  FLACC scale will be measured as following:
  Each category (face,legs,activity, and cry consolability) is scored on the 0-2 scale which results in a total score of 0-10.
  Assessment of the final score:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain

SECONDARY OUTCOMES:
pain scores | at 2 hour intervals during the first 24 hours postoperatively
  By using face, legs, activity, and cry consolability scale [FLACC ]
  FLACC scale will be measured as following:
  Each category (face,legs,activity, and cry consolability) is scored on the 0-2 scale which results in a total score of 0-10.
  Assessment of the final score:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Block failure rate | First hour postoperatively
  The block will be considered a failed block if the patient required more than two doses of rescue analgesia in the first hour postoperatively
Block performance time | Preoperative
The incidence of adverse effects | Up to one week after the block
Duration of the block | UP to 48 hours postoperatively
Degree of contralateral motor blockage and lower limb weakness | UP to 48 hours postoperatively
  By using modified bromage scale as following:
  Grade I : Free movement of legs and feet Degree of block :Nil (0%)
  Grade II :Just able to flex knees with free movement of feet Degree of block :Partial (33%)
  Grade III :Unable to flex knees, but with free movement of feet Degree of block: Almost complete (66%)
  Grade IV :Unable to move legs or feet Degree of block: Complete (100%)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini hospital, Cairo, Egypt